CLINICAL TRIAL: NCT05571150
Title: A Novel Rehabilitation Approach for Optimizing Dyadic Outcomes of Stroke Survivors and Their Caregivers: Dyadic Strategy Training
Brief Title: A Novel Rehabilitation Approach: Dyadic Strategy Training for Stroke Survivors and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Feng-Hang Chang, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202203083
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention group (Experimental): The dyad-focused strategy training intervention will be delivered to the treatment group. The intervention protocols of the dyad-focused strategy training were developed based on the strategy training guideline outlined by Skidmore et al, Bodenmann's framework of dyadic coping, and the self-efficacy theory.
  Interventions: Behavioral: Dyad-focused strategy training intervention
- Control intervention group (Active Comparator): Participants in the control group will receive a dose-matched stroke education provided by a trained research therapist as an attention-control intervention. The therapist will provide in-person education to the dyad using an illustrated manual developed based on the stroke rehabilitation guidelines suggested by the American Heart Association/American Stroke Association .
  Interventions: Behavioral: Attention-control intervention

INTERVENTIONS:
Behavioral: Dyad-focused strategy training intervention — The program consists of five critical ingredients: shared decision making, self-selected goals, self-evaluation of performance, strategy development and implementation, and therapeutic guided discovery.
  Trained research therapists will deliver the intervention to the survivor-caregiver dyads on a one-to-two base at the participants' home or in a quiet room at our collaborative hospitals. The therapist will ask the dyad to identify 3 to 5 shared participation goals and provide them the global strategy (also called guided discovery strategy), which involves (1) setting a goal to address the barriers, (2) developing a plan to address the goal, (3) doing the plan, and (4) checking if the plan worked or required revising. This procedure will be repeated iteratively until the dyad's goal is met, and the next goal can be moved on to.
  Arms: Experimental intervention group
Behavioral: Attention-control intervention — The topics of the education will cover: (1) secondary stroke prevention; (2) prevention and management of comorbidities; (3) managing emotions and behaviors; (3) medications and personal care; (4) finances and transportation; and (5) home and community-based participation.
  Arms: Control intervention group

SUMMARY:
The purpose of this study is to examine the efficacy of a newly developed dyad-focused strategy training intervention on enhancing participation of stroke survivors and their caregivers.

To address this purpose, a single-blinded, parallel-group randomized controlled trial will be implemented to assess the efficacy of the dyad-focused strategy training intervention in comparison to the control group. An expected sample of 138 stroke survivor-caregiver dyads will be recruited from our collaborative hospitals in Northern Taiwan.

Data will be analyzed using multiple linear regression models and mixed-effects regression models. Qualitative in-depth interviews with participants, caregivers, and therapists will be conducted following the intervention.

Findings of this study will provide important evidence on whether this newly-developed program has immediate and long-term effect on improving and maintaining participation for both stroke survivors and their caregivers. These findings will together support the application of the dyad-focused strategy training intervention in rehabilitation practice and inform future study development.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and adult disability. Stroke survivors and their caregivers often experience an overwhelming sense of social isolation and experience a wide range of participation restrictions after stroke, leading to frustration and adverse health outcomes. To address both the survivor and caregiver needs, dyad-focused interventions are necessary to be implemented in the transitioning process. However, very few interventions were designed to address the needs of the dyad and place an equal emphasis on both survivors' and caregivers' outcomes. The purpose of this study is to examine the efficacy of a newly developed dyad-focused strategy training intervention on enhancing participation of stroke survivors and their caregivers.

To address this purpose, a single-blinded, parallel-group randomized controlled trial will be implemented to assess the efficacy of the dyad-focused strategy training intervention in comparison to the control group. An expected sample of 138 stroke survivor-caregiver dyads will be recruited from our collaborative hospitals in Northern Taiwan. These participants will be randomly assigned to the intervention group and the control group at a 1:1 ratio. Outcome measures including the Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D), General Self-Efficacy Scale (GSES), Activity Measure for Post-Acute Care (AM-PAC), and other standardized assessment tools and questionnaires will be administered to the participants at baseline (T1), post-intervention (T2), and 3-month (T3), and 6-month (T4) follow-ups. Data will be analyzed using multiple linear regression models and mixed-effects regression models.

Qualitative in-depth interviews with participants, caregivers, and therapists will be conducted following the intervention. Data regarding the interviewees' experiences, satisfaction, and their perceived effectiveness of the intervention will be collected. Transcribed data will be coded by two independent coders and analyzed with thematic analysis method.

Findings of this study will provide important evidence on whether this newly-developed program has immediate and long-term effect on improving and maintaining participation for both stroke survivors and their caregivers. The mechanism of whether and how this intervention program impacts the dyad's self-efficacy and the functions of stroke survivors in addition to participation will also be identified. These findings will together support the application of the dyad-focused strategy training intervention in rehabilitation practice and inform future study development.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors

  1. ages 20 years and older;
  2. has been diagnosed with a first-time stroke within the past two year;
  3. speaks Mandarin;
  4. has an identified primary caregiver who provides care or assistance of any kind and taking responsibility for the survivor;
  5. is able to provide informed consent.
* Family caregivers include that the caregiver

  1. ages 20 years and older;
  2. speaks Mandarin;
  3. is the primary caregiver recognized by the survivor;
  4. is available to participate in the intervention sessions with the survivor;
  5. is able to provide informed consent.

Exclusion Criteria:

* The survivor-caregiver dyad will be excluded if any of them:

  1. requires significant medical treatment (e.g., chemotherapy, radiation therapy, or hemo/peritoneal dialysis) that may impede them from participating in the study;
  2. has severe aphasia;
  3. is unable to participate in a 1-hour discussion session;
  4. has a diagnosis of dementia, major depressive disorder, substance use or other psychiatric disorders that may impede them from participating in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to up to 6 weeks
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.

SECONDARY OUTCOMES:
World Health Organization Quality of Life (WHOQOL-Brief) | From baseline to up to 6 weeks
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
World Health Organization Quality of Life (WHOQOL-Brief) | From baseline to up to 18 weeks
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
World Health Organization Quality of Life (WHOQOL-Brief) | From baseline to up to 30 weeks
  The WHOQOL-BREF (Taiwan ver.) is a self-administered questionnaire comprising 28 questions on individuals' perceptions of their health and well-being over the previous two weeks. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely".
General Self-Efficacy Scale (GSES) | From baseline to up to 6 weeks
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
General Self-Efficacy Scale (GSES) | From baseline to up to 18 weeks
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
General Self-Efficacy Scale (GSES) | From baseline to up to 30 weeks
  The GSES, sometimes seen as GSE, is a 10-item psychometric scale created to assess perceived self-efficacy regarding coping and adaptation abilities in daily activities and isolated stressful events. Responses to questions are on a 1-4 Likert scale where 1 represents "Not at all true" and 4 represents "Exactly true."
Activity Measure for Post-Acute Care (AM-PAC) Short Forms | From baseline to up to 6 weeks
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AM-PAC) Short Forms | From baseline to up to 18 weeks
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Activity Measure for Post-Acute Care (AM-PAC) Short Forms | From baseline to up to 30 weeks
  The AM-PAC consists of three subscales that assess three activity domains: basic mobility, daily activity, and applied cognitive. The inpatient short consists of 6 items per domain, and the outpatient short consists of 15-19 per domain. Each item asks the respondent to rate the difficulty of performing specified activities using a 4-point scale. The summary scores for each subscale will be transformed into standardized scores on the t-score scale.
Montreal Cognitive Assessment (MoCA) | From baseline to up to 6 weeks
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Montreal Cognitive Assessment (MoCA) | From baseline to up to 18 weeks
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Montreal Cognitive Assessment (MoCA) | From baseline to up to 30 weeks
  MoCA is a 30-question test. It checks different cognitive or thinking abilities to help people quickly assess a patient's cognitive health.
  The score ranges from 0 to 30. A score of 26 and higher is considered normal.
Stroop Test | From baseline to up to 6 weeks
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
Stroop Test | From baseline to up to 18 weeks
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
Stroop Test | From baseline to up to 30 weeks
  The Stroop test assesses the ability to inhibit cognitive interference that occurs when processing a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute. Participants will be asked to read out the word's ink color as accurately as soon as possible. The ink color of the word could be congruent or incongruent with the written color name. Each participant's time to complete the task will be calculated and recorded.
TMT Test | From baseline to up to 6 weeks
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking.
TMT Test | From baseline to up to 18 weeks
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking.
TMT Test | From baseline to up to 30 weeks
  The TMT test measures sustained attention, sequencing, mental flexibility, and visual tracking.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to up to 18 weeks
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.
Participation Measure- 3 Domains, 4 Dimensions (PM-3D4D) | From baseline to up to 30 weeks
  The PM-3D4D is a 24-item measure that was designed to evaluate three domains of participation: Productivity, Social, and Community.

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Hang Chang, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin YN, Hsu SP, Kang JH, Liou TH, Han DS, Ni P, Chiu V, Rodakowski J, Chang FH. Enhancing dyadic outcomes of stroke survivors and caregivers: protocol for a randomised controlled trial. BMJ Open. 2025 May 21;15(5):e090751. doi: 10.1136/bmjopen-2024-090751. PMID 40398954